CLINICAL TRIAL: NCT00800514
Title: Amantadine and Temporal Discrimination in Patients With Traumatic Brain Injury
Brief Title: Amantadine and Temporal Discrimination in Patients With Traumatic Brain Injury (TBI)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator took a position at another institution. No subjects enrolled.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 08-01
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-02

CONDITIONS: Traumatic Brain Injury
Keywords: perception of time, traumatic brain injury, amantadine
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- active (Experimental)
  Interventions: Drug: amantadine

INTERVENTIONS:
Drug: amantadine — amantadine twice daily
Drug: amantadine — amantadine 100 mg twice daily

SUMMARY:
The study will explore the neurocognitive effect of four weeks of treatment with amantadine versus placebo in patients with traumatic brain injury using the Interval Bisection Timing Task. Approximately 16 individuals with traumatic brain injury are expected to participate in this study. Subject participation is expected to last up to 8 weeks with 16 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 inclusive. History of post-MVA close head TBI. Female subjects must use an acceptable method of contraception during entire study. Acceptable methods of contraception are: history of surgical sterility, postmenopausal status, hormonal contraceptives, or accepted barrier devices (i.e., male/female condom, diaphragm, cervical cap, intrauterine device).

Exclusion Criteria:

* Current or past history of major psychiatric disorder (schizophrenia, bipolar disorder, major depressive disorder)
* Substance use disorder
* Current or past history of serious chronic medical condition (pulmonary (lung), cardiovascular (heart), hepato-renal (liver-kidney) disease, diabetes)
* Seizures
* Smoking one or more packs of cigarettes per day
* If you are pregnant or breastfeeding, or plan to become pregnant during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the Interval Bisection Timing Task. | 12 -16 months

SECONDARY OUTCOMES:
The secondary efficacy measure is the Barrett Impulsiveness Scale (BIS-11). | 12-16 moths

CONTACTS AND LOCATIONS:
Overall Officials: Oleg V. Tcheremissine, MD, Principal Investigator — Carolians HealthCare System
Locations (1):
- CHS-Behavioral Health Research, Charlotte, North Carolina, United States

REFERENCES:
- See also: Click here for more information about this study and CHS — http://www.carolinashealthcare.org